### STATISTICAL ANALYSIS PLAN -- MOCK UP DISPLAYS

Title: An Open-Label Safety, Tolerability, and Efficacy Study in Male and Female Subjects with Androgenetic Alopecia Treated with ATI-50002 Topical Solution

Protocol:

ATI-50002-AGA-201

Study Drug: ATI-50002

Sponsor:

Aclaris Therapeutics, Inc.

Date:

23-April 2019

Status:

Final 1.0

Prepared by:

John Ilgenfritz: Statistical Consultant

Approved by:

Aclaris:

David Burt: Sr. Director, Biostatistics

Date: 23 Mar 2019

## **END-OF-TEXT TABLES**

| Number | Title |
|---|---|
| Table 14.1.1.1 | Study Population and Patient Disposition |
| Table 14.1.1.2 | Reasons for Discontinuation from Study ITT Population |
| Table 14.1.2 | Patient Demographics and Other Baseline Characteristics ITT Population |
| Table 14.1.3 | Diagnosis and Prior Treatments for Androgenetic Alopecia Safety |
| | Population |
| Table 14.1.4 | Exposure to Study Medication Safety Population |
| Table 14.1.5 | Exposure to Study Medication Safety Population |
| Table 14.2.1.1 | Non-Vellus Target Area Hair Count (TAHC): Mean and Mean Change |
| | from Baseline (hairs/cm <sup>2</sup> ) ITT Population |
| Table 14.2.1.2 | Vellus Target Area Hair Count: Mean and Mean Change from Baseline |
| | (hairs/cm <sup>2</sup> ) ITT Population |
| Table 14.2.1.3 | Total (Non-Vellus + Vellus) Target Area Hair Count: Mean and Mean |
| | Change from Baseline (hairs/cm <sup>2</sup> ) ITT Population |
| Table 14.2.1.4 | Non-Vellus Target Area Hair Width: Mean and Mean Change from |
| | Baseline (cm) ITT Population |
| Table 14.2.1.5 | Vellus Target Area Hair Width: Mean and Mean Change from Baseline |
| | (cm) ITT Population |
| Table 14.2.1.6 | Total (Non-Vellus + Vellus) Target Area Hair Width: Mean and Mean |
| | Change from Baseline (cm) ITT Population |
| Table 14.2.1.7 | Average Non-Vellus Hair Width: Mean and Mean Change from Baseline |
| | (cm) ITT Population |
| Table 14.2.2.1 | Investigator Global Assessment ITT Population |
| Table 14.2.2.2 | Subject Self-Assessment ITT Population |
| Table 14.2.3.1 | Investigator Global Assessment: Patients with Slightly Increased Hair |
| | Growth or Better (Grade +1 to +3) ITT Population |
| Table 14.2.3.2 | Subject Self-Assessment: Patients with Slightly Increased Hair Growth or |
| | Better (Grade +1 to +3) ITT Population |
| Table 14.2.4 | Improvement from Baseline in Norwood-Hamilton Scale in Males ITT |
| | Population |
| Table 14.2.5 | Improvement from Baseline in Sinclair Scale in Females Safety |
| | Population |
| Table 14.2.6 | Correlation of Selected Effiacy Measures ITT Population |
| Table 14.2.7 | Correlation of Nonvellus Hair Count and Width Measures with Time |
| | Since Diagnosis of Androgenetic Alopecia ITT Population |
| Table 14.3.1 | Summary of Treatment-Emergent Adverse Events Safety Population |
| Table 14.3.1.1 | Treatment-Emergent Adverse Events by System Organ Class and |
| T 11 14010 | Preferred Term Safety Population |
| Table 14.3.1.2 | Treatment-Emergent Study Treatment-Related Adverse Events by System |
| T 11 14212 | Organ Class and Preferred Term Safety Population |
| Table 14.3.1.3 | Treatment-Emergent Adverse Events Resulting in Discontinuation of |
| | Study Treatment by System Organ Class and Preferred Term Safety |
| | Population |

| Table 14.3.1.4 | Treatment-Emergent Serious Adverse Events by System Organ Class and Preferred Term Safety Population |
|---|---|
| Table 14.3.1.5 | Treatment-Emergent Adverse Events by Descending Order of Frequency for ATI-50002 Safety Population |
| Table 14.3.1.6 | Treatment-Emergent Adverse Events by Maximum Severity Safety Population |
| Table 14.3.1.7 | Treatment-Emergent Study Medication Related Adverse Events by Maximum Severity Safety Population |
| Table 14.3.1.8 Safety Population | Local Skin Reactions – Highest Grade Any Time Post-Baseline |
| Table 14.3.1.9 | Treatment-Emergent Adverse Events by System Organ Class and<br>Preferred Term in Patients Who Discontinued in First 26 Weeks Safety<br>Population |
| Table 14.3.1.10 | Treatment-Emergent Adverse Events by System Organ Class and Preferred Term in Patients Who Completed 26 Weeks and Did not Enter Six Month Extension Safety Population |
| Table 14.3.1.11 | Treatment-Emergent Adverse Events by System Organ Class and Preferred Term in Patients Who Completed 26 Weeks and Entered Six Month Extension Safety Population |
| Table 14.3.2.1 | Vital Signs: Systolic Blood Pressure (mmHg) Safety Population |
| Table 14.3.2.2 | Vital Signs: Diastolic Blood Pressure (mmHg) Safety Population |
| Table 14.3.2.3 | Vital Signs: Heart Rate (bpm) Safety Population |
| Table 14.3.2.4 | Vital Signs: Respiratory Rate (bpm) Safety Population |
| Table 14.3.2.5 | Vital Signs: Temperature (Degrees C) Safety Population |
| Table 14.3.3 | ECG Interpretation: Shift from Baseline to Worst Assessment Post |
| Table 14.3.4.1 | Baseline Safety Population Descriptive Statistics for Chamistry Population |
| Table 14.3.4.1 Table 14.3.4.2 | Descriptive Statistics for Chemistry Parameters Safety Population Descriptive Statistics for Hematology Parameters Safety Population |
| Table 14.3.4.3 | Descriptive Statistics for Hernatology Farameters Safety Population |
| Table 14.3.5 | Number and Percent of Patients Meeting Criteria for Hepatobiliary |
| 14010 17.3.3 | Laboratory Abnormalities Safety Population |
| Table 14.3.6 | Number and Percent of Patients Meeting Laboratory Criteria for Potential Renal Impairment Safety Population |

Aclaris Therapeutics Inc.
Protocol: ATI-50002-AGA-201

## **END-OF-TEXT FIGURES**

| Number | <u>Title</u> |
|---|---|
| Figure 14.1 | Association of Selected Efficacy Measures with Fit Linear Regression Line |
| Figure 14.2 | Association of Selected Efficacy Measures with Fit Linear Regression Line, ITT Population: Visit=V7 Week 16 |
| Figure 14.3 | Association of Selected Efficacy Measures with Fit Linear Regression Line, ITT Population: Visit=V10 Week 26 |
| Figure 14.4 | Association of Selected Efficacy Measures with Fit Linear Regression Line, ITT Population: Visit=V16 Week 52 |
| Figure 14.5 | Association of Change in Nonvellus Target Area Average Hair Width with Investigator Global Assessment, ITT Population |
| Figure 14.6 | Association of Change in Nonvellus Target Area Average Hair Width with Subject Self Assessment, ITT Population |
| Figure 14.7 | Association of Change in Nonvellus Target Area Hair Count with Time Since Diagnosis of Androgenetic Alopecia, ITT Population |
| Figure 14.8 | Association of Change in Nonvellus Target Area Hair Width with Time Since Diagnosis of Androgenetic Alopecia, ITT Population |
| Figure 14.9 | Association of Change in Nonvellus Target AreaAverage Hair Width with Time Since Diagnosis of Androgenetic Alopecia, ITT Population |

## PATIENT DATA LISTINGS

| Number | <u>Title</u> |
|---|---|
| Appendix 16.2.1.1 | Disposition |
| Appendix 16.2.1.2 | Demographics |
| Appendix 16.2.1.3 | History of Androgenetic Alopecia: Diagnosis and Prior Treatment and |
| | Therapies |
| Appendix 16.2.1.4 | Medical History |
| Appendix 16.2.1.5 | Prior and Concomitant Therapies |
| Appendix 16.2.1.6 | ATI-50002 Accountability |
| Appendix 16.2.1.7 | ATI-50002 Accountability Comments |
| Appendix 16.2.1.8 | ATI-50002 Application Changes and Missed Doses |
| Appendix 16.2.1.9 | Eligibility Criteria |
| Appendix 16.2.1.10 | Protocol Violations |
| Appendix 16.2.2.1 | Target Area Hair Count and Width |
| Appendix 16.2.2.2 | Investigator and Subject Global Assessments |
| Appendix 16.2.2.3 | Norwood-Hamilton Scale in Males |
| Appendix 16.2.2.4 | Sinclair Scale in Females |
| Appendix 16.2.3.1 | All Adverse Events |
| Appendix 16.2.3.2 | Serious Adverse Events |
| Appendix 16.2.3.3 | Adverse Events Resulting in Discontinuation of Study Treatment |
| Appendix 16.2.3.4 | Adverse Events Resulting in Outcome of Death |
| Appendix 16.2.3.5 | Local Skin Reactions |
| Appendix 16.2.3.6 | Physical Exam |
| Appendix 16.2.3.7 | Vital Signs |
| Appendix 16.2.3.8 | Electrocardiogram – Evaluator Interpretation |
| Appendix 16.2.3.9 | Clinical Laboratory Assessments: Hematology |
| Appendix 16.2.3.10 | Clinical Laboratory Assessments: Biochemistry |
| Appendix 16.2.3.11 | Clinical Laboratory Assessments: Hormones |
| Appendix 16.2.3.12 | Clinical Laboratory Assessments: Urinalysis |
| Appendix A | MedDRA System Organ Class/Preferred Term and CRF Verbatim Terms |

# MOCKUPS OF TABLES, AND PATIENT LISTINGS

Aclaris Therapeutics Inc.

23 Apr 2019 Statistical Analysis Plan

Protocol: ATI-50002-AGA-201

**Table 14.1.1.1 Study Population and Patient Disposition** 

| | Female<br>n (%) | Male<br>n (%) | Total<br>n (%) |
|---|---|---|---|
| Population/Group | | | |
| Intent-to-Treat (ITT) Population | xx (100) | xx (100 | xx (100 |
| Safety Population | xx (100) | xx (100 | xx (100 |
| Entered 6 Month Extension | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: Percentages based on the number of patients receiving at least 1 treatment application

Table 14.1.1.2
Reasons for Discontinuation from Study
ITT Population

| | Female<br>(N=xxx) | Male<br>(N=xxx) | Total (N=xxx) |
|---|---|---|---|
| | n (%) | n (%) | n (%) |
| ENTIRE STUDY <sup>a</sup> : | | | |
| Number (%) of Patients Discontinued | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Protocol Violation | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| AE/SAE | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Lost to Follow-Up | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Withdrew Consent | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Pregnancy | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| Other | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| Completed 26 Week Study | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| Completed Optional 6 Month Extension | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| Ongoing as of "cut-off date" | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| FIRST 26 WEEKS: | | | |
| Number (%) of Patients Discontinued | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Protocol Violation | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| AE/SAE | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| Lost to Follow-Up | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| Withdrew Consent | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| Pregnancy | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| Other | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| Completed | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| Ongoing as of "cut-off date" | xx(xx.x) | xx (xx.x) | xx (xx.x) |

<sup>&</sup>lt;sup>a</sup> Includes all discontinuations/completions from the first 26 weeks and optional 6 month extension. Patents completing both the initial 26 weeks and the 6 month extension periods are counted on both corresponding rows.

<sup>&</sup>lt;sup>b</sup> Used as denominator for percentages calculated under 6 month extension.

Table 14.1.1.2
Reasons for Discontinuation from Study
ITTSafety Population

| | Female<br>(N=xxx)<br>n (%) | Male<br>(N=xxx)<br>n (%) | Total<br>(N=xxx)<br>n (%) |
|---|---|---|---|
| 6 MONTH EXTENSION: | | | |
| Number of Patients Entering <sup>b</sup> | xx | XX | xx |
| Number (%) of Patients Discontinued | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Protocol Violation | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| AE/SAE | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to Follow-Up | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| Withdrew Consent | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| Pregnancy | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| Completed | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| Ongoing as of "cut-off date" | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>&</sup>lt;sup>a</sup> Includes all discontinuations/completions from the first 26 weeks and optional 6 month extension. Patents completing both the initial 26 weeks and the 6 month extension periods are counted on both corresponding rows.

<sup>&</sup>lt;sup>b</sup> Used as denominator for percentages calculated under 6 month extension.

Table 14.1.2
Patient Demographics and Other Baseline Characteristics
ITT Population

| | Female | Male | Total |
|---|---|---|---|
| | (N=xxx) | (N=xxx) | (N=xxx) |
| Age (years) | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | XX.X | XX.X |
| Min, Max | XX,XX | XX,XX | XX,XX |
| Age Category (years), n (%) | | | |
| < 35 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ≥ 35 | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Gender, n (%) | | | |
| Male | | | xx (xx.x) |
| Female | | | xx(xx.x) |
| Race, n (%) | | | |
| White | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Black or African American | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Asian | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| American Indian or Alaska Native | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Native Hawaiian or Other Pacific Islander | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ethnicity, n (%) | | | |
| Hispanic or Latino | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Non-Hispanic or Latino | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Reported | ` / | ` / | ` / |

Table 14.1.2
Patient Demographics and Other Baseline Characteristics
ITT Population

| | Female | Male | Total |
|--------------------------------|-----------|-----------|-----------|
| | (N=xxx) | (N=xxx) | (N=xxx) |
| Height (cm) | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX |
| Weight (kg) | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | xx, xx |
| Fitzpatrick Skin Type, n (%) | | | |
| 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4 | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| 5 | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| 6 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Sinclar Grade (Females), n (%) | | | |
| 2 | xx(xx.x) | | |
| 3 | xx (xx.x) | | |
| 4 | xx(xx.x) | | |

Table 14.1.2
Patient Demographics and Other Baseline Characteristics
ITT Population

| | Female<br>(N=xxx) | Male<br>(N=xxx) | Total<br>(N=xxx) |
|---|---|---|---|
| Norwood-Hamilton Classificiation (Males), n (%) | | | |
| III vertex | | xx (xx.x) | |
| IV | | xx (xx.x) | |
| IVa | | xx (xx.x) | |
| | | xx (xx.x) | |

Table 14.1.3
Diagnosis and Prior Treatments for Androgenetic Alopecia
Safety Population

| | Female | Male | Total |
|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) |
| Prior Therapies for Androgenetic Alopecia, n (%) | | | |
| ANY therapy | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| Minoxidil | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| Finasteride | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Device | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| {Will need to review for appropriate categories} | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Fime since Diagnosis of Androgenetic Alopecia (Weeks) <sup>a</sup> | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx |
| Age at Diagnosis of Androgenetic Alopecia (Years) | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX |

<sup>&</sup>lt;sup>a</sup> (date of first application of study medication – date of diagnosis)/7.

Table 14.1.4 Exposure to Study Medication Safety Population

| | Female | Male | Total |
|--------------------------------------------|--------|--------|--------|
| Parameter | (N=xx) | (N=xx) | (N=xx) |
| Duration of Treatment (Weeks) <sup>a</sup> | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx |
| Total Weight Administered (gm) | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | xx.xx | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx |
| Total Volume Administered (mL) | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | xx.xx | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | xx, xx |

 $<sup>^{</sup>a}$  (Date of last application of study medication – date of first application of study medication +1 ) / 7. Includes exposure in optional six month extension, if applicable.

<sup>&</sup>lt;sup>b</sup> Each patient's average volume across all applications is calculated first.

Table 14.1.5 Exposure to Study Medication Safety Population

| | Female | Male | Total |
|---|---|---|---|
| Parameter | (N=xx) | (N=xx) | (N=xx |
| Fotal Number of Applications (Total of Each Patient | t) | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | xx.xx | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX |
| Total Applications (All Patients Total) | XXXX | XXXX | XXXX |
| Average Volume Per Application (mL) <sup>b</sup> | | | |
| N | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | xx.xx | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX |

<sup>&</sup>lt;sup>a</sup> (Date of last application of study medication – date of first application of study medication +1) / 7. Includes exposure in optional six month extension, if applicable.

<sup>&</sup>lt;sup>b</sup> Each patient's average volume across all applications is calculated first.

23 Apr 2019 Statistical Analysis Plan

**Table 14.2.1.1** Non-Vellus Target Area Hair Count (TAHC): Mean and Mean Change from Baseline (hairs/cm²) **ITT Population** 

| | | Fen | nale | Male | | To | otal |
|---|---|---|---|---|---|---|---|
| Visit | Statistic | Value | Change | Value | Change | Value | Change |
| D 1' a | | | | | | | |
| Baseline <sup>a</sup> | n | XX | | XX | | XX | |
| | Mean (SD) | xx.x(xx.xx) | | xx.x (xx.xx) | | xx.x(xx.xx) | |
| | SE | X.XX | | X.XX | | X.XX | |
| | Median | XXX.X | | XXX.X | | XXX.X | |
| | (Min, Max) | (xxx, xxx) | | (xxx,xxx) | | (xxx,xxx) | |
| V5 – Week 8 | n | XX | XX | XX | XX | XX | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | SÈ | x.xx | X.XX | X.XX | x.xx | x.xx | x.xx |
| | Median | XXX.X | XXX.X | XXX.X | xxx.x | XXX.X | XXX.X |
| | (Min, Max) | (xxx,xxx) | (xxx, xxx) | (xxx,xxx) | (xxx,xxx) | (xxx,xxx) | (xxx,xxx) |
| | [95% CI] <sup>b</sup> | () | [xx.x, xx.x] | ( ,) | [xx.x, xx.x] | ( ;) | [xx.x, xx.x] |
| V7– Week 16 | n | XX | XX | XX | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | SE | x.xx | X.XX | X.XX | x.xx | X.XX | x.xx |
| | Median | XXX.X | XXX.X | XXX.X | xxx.x | XXX.X | xxx.x |
| | (Min, Max) | (xxx,xxx) | (xxx,xxx) | (xxx,xxx) | (xxx, xxx) | (xxx,xxx) | (xxx, xxx) |
| | [95% CI] <sup>b</sup> | ()) | [xx.x, xx.x] | () | [xx.x, xx.x] | () | [xx.x, xx.x] |

 <sup>&</sup>lt;sup>a</sup> Baseline is selected as the last measurement prior to the first application of study medication.
 <sup>b</sup> Confidence interval for the change from baseline.

Protocol: ATI-50002-AGA-201

Table 14.2.1.1 Non-Vellus Target Area Hair Count: Mean and Mean Change from Baseline (hairs/cm²) ITT Population

| | | Fen | nale | Ma | ale | To | tal |
|---|---|---|---|---|---|---|---|
| Visit | Statistic | Value | Change | Value | Change | Value | Change |
| V10-Week 26 | n<br>Mean (SD)<br>SE<br>Median<br>(Min, Max)<br>[95% CI] <sup>b</sup> | xx<br>xx.x (xx.xx)<br>x.xx<br>xxx.x<br>(xxx ,xxx) | XX XX.X (XX.XX) X.XX XXX.X (XXX ,XXX) | xx<br>xx.x (xx.xx)<br>x.xx<br>xxx.x<br>(xxx ,xxx) | XX XX.X (XX.XX) X.XX XXX.X (XXX, XXX) | xx<br>xx.x (xx.xx)<br>x.xx<br>xxx.x<br>(xxx ,xxx) | XX XX.X (XX.XX) X.XX XXX.X (XXX, XXX) |
| V16-Week 52 | n<br>Mean (SD)<br>SE<br>Median<br>(Min, Max)<br>[95% CI] <sup>b</sup> | xx<br>xx.x (xx.xx)<br>x.xx<br>xxx.x<br>(xxx ,xxx) | [xx.x, xx.x] xx xx.x (xx.xx) x.xx xxx.x (xxx, xxxx) [xx.x, xx.x] | xx<br>xx.x (xx.xx)<br>x.xx<br>xxx.x<br>(xxx ,xxx) | [xx.x, xx.x] xx xx.x (xx.xx) x.xx xxx.x (xxx, xxxx) [xx.x, xxxx) | xx<br>xx.x (xx.xx)<br>x.xx<br>xxx.x<br>(xxx ,xxx) | [xx.x, xx.x] xx xx.x (xx.xx) x.xx xxx.x (xxx, xxxx) [xx.x, xx.x] |

<sup>&</sup>lt;sup>a</sup> Baseline is selected as the last measurement prior to the first application of study medication.

#### Repeat Format for

Table 14.2.1.2 Vellus Target Area Hair Count: Mean and Mean Change from Baseline (hairs/cm²) ITT Population

Table 14.2.1.3 Total (Non-Vellus + Vellus) Target Area Hair Count: Mean and Mean Change from Baseline (hairs/cm²) ITT Population

Table 14.2.1.4 Non-Vellus Target Area Hair Width: Mean and Mean Change from Baseline (cm) ITT Population

Table 14.2.1.5 Vellus Target Area Hair Width: Mean and Mean Change from Baseline (cm) ITT Population

Table 14.2.1.6 Total (Non-Vellus + Vellus) Target Area Hair Width: Mean and Mean Change from Baseline (cm) ITT Population

 Table 14.2.1.7
 Average Non-Vellus Hair Width: Mean and Mean Change from Baseline (cm) ITT Population

Footnote for 14.2.1.7: Note: Average non-vellus hair width is calculated for each patient as the non-vellus target area count divided by the non-vellus target area hair width

<sup>&</sup>lt;sup>b</sup> Confidence interval for the change from baseline.

23 Apr 2019 Statistical Analysis Plan

Table 14.2.2.1 Investigator Global Assessment ITT Population

| | | ITT Population | | |
|---|---|---|---|---|
| Visit | Statistic | Female | Male | Total |
| V5 – Week 8 | n | XX | XX | VV |
| v 5 – vv eek o | Mean (SD) | | | XX |
| | ` , | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xxx.x | XXX.X | XXX.X |
| | (Min, Max) | (xxx,xxx) | (xxx,xxx) | (xxx, xxx) |
| V7– Week 16 | n | XX | xx | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xxx.x | XXX.X | XXX.X |
| | (Min, Max) | (xxx,xxx) | (xxx,xxx) | (xxx,xxx) |
| V10-Week 26 | n | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XXX.X | XXX.X | XXX.X |
| | (Min, Max) | (xxx, xxx) | (xxx, xxx) | (xxx, xxx) |
| V13-Week 39 | n | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XXX.X | XXX.X | XXX.X |
| | (Min, Max) | (xxx,xxx) | (xxx,xxx) | (xxx,xxx) |
| V16 – Week 52 | n | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x(xx.xx) | xx.x(xx.xx) |
| | Median | XXX.X | XXX.X | XXX.X |
| | (Min, Max) | (xxx, xxx) | (xxx, xxx) | (xxx, xxx) |
| FU/Early Termination | n | XX | XX | XX |
| 1 C. Larry 1 Crimmunon | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XXX.X | XXX.X | XXX.X |
| | (Min, Max) | | | |
| | (IVIIII, IVIAX) | (xxx ,xxx) | (xxx ,xxx) | (xxx, xxx) |

Repeat Format for

 Table 14.2.2.2
 Subject Self-Assessment ITT Population

Aclaris Therapeutics Inc.

Protocol: ATI-50002-AGA-201

23 Apr 2019 Statistical Analysis Plan

Table 14.2.3.1
Investigator Global Assessment: Patients with Slightly Increased Hair Growth or Better (Grade +1 to +3)
ITT Population

| Visit | Statistic | Female | Male | Total |
|---|---|---|---|---|
| V5 – Week 8 | $N^a$ n (%) | xx xx (xx.x) | xx xx (xx.x) | xx xx (xx.x) |
| V7- Week 16 | $N^a$ n (%) | xx xx (xx.x) | xx xx (xx.x) | xx xx (xx.x) |
| V10-Week 26 | $N^a$ n (%) | xx xx (xx.x) | xx xx (xx.x) | xx xx (xx.x) |
| V13-Week 39 | $N^a$ n (%) | xx xx (xx.x) | xx xx (xx.x) | xx xx (xx.x) |
| V16 – Week 52 | $N^a$ n (%) | xx xx (xx.x) | xx xx (xx.x) | xx xx (xx.x) |
| FU/Early Termination | $N^a$ n (%) | xx xx (xx.x) | xx xx (xx.x) | xx xx (xx.x) |

### **Repeat Format for**

Table 14.2.3.2 Subject Self-Assessment: Patients with Slightly Increased Hair Growth or Better (Grade +1 to +3) ITT Population

<sup>&</sup>lt;sup>a</sup> The number of patents with an assessement at the visit. Used as denominator for percentages.

Table 14.2.4
Improvement from Baseline in Norwood-Hamilton Scale in Males
ITT Population

| Visit | = | Improved by $\geq 1$ Level | Improved by $\geq 2$ Levels |
|---|---|---|---|
| Shift Detail <sup>a</sup> | $N^b$ | n (%) | n (%) |
| V7 – Week 16 | XX | xx (xx.x) | xx(xx.x) |
| IV – IIIa | | xx (xx.x) | xx (xx.x) |
| IV – III vertex | | xx (xx.x) | |
| etc | | | |
| V10 – Week 26 | XX | xx (xx.x) | xx (xx.x) |
| IV – IIIa | | xx (xx.x) | xx (xx.x) |
| IV – III vertex | | xx (xx.x) | |
| etc | | | |
| V16 – Week 52 | XX | xx (xx.x) | xx (xx.x) |
| IV – IIIa | | xx (xx.x) | xx (xx.x) |
| IV – III vertex | | xx (xx.x) | , , |
| etc | | ` ' | |
| FU/Early Termination <sup>c</sup> | XX | xx (xx.x) | xx (xx.x) |
| IV – IIIa | | xx (xx.x) | xx (xx.x) |
| IV – III vertex | | xx (xx.x) | , |
| etc | | , | |
| Early Term, 1st 26 Weeks | XX | xx (xx.x) | xx (xx.x) |
| IV – IIIa | | xx (xx.x) | xx (xx.x) |
| IV – III vertex | | xx (xx.x) | 9 |
| etc | | ini (mini) | |

 $<sup>^{</sup>a}$  The Baseline Score →Timepoint Score combination that met the ≥ 1 level improvement criteria.

<sup>&</sup>lt;sup>b</sup> The number of patients with a non-missing score baseline and at the visit indicated. Used as denominator for percentages.

<sup>&</sup>lt;sup>c</sup> Includes early terminations or follow-ups collected during the first 26 Weeks or during the additional six months for patients opting to continue treatment in the optional six month extension. Additional rows provided to further sub-divide based on the period (1<sup>st</sup> 26 Weeks vs 6 Month Extension) and termination status (early termination vs follow-up).

Protocol: ATI-50002-AGA-201

Table 14.2.4
Improvement from Baseline in Norwood-Hamilton Scale in Males
ITT Population

| Visit<br>Shift Detail <sup>a</sup> | $N^b$ | Improved by ≥ 1 Level n (%) | Improved by $\geq 2$ Levels n (%) |
|---|---|---|---|
| E II 4st AC W | | () | () |
| Follow-Up 1st 26 Weeks | XX | xx (xx.x) | xx(xx.x) |
| IV – IIIa | | xx (xx.x) | xx(xx.x) |
| IV – III vertex | | xx (xx.x) | |
| etc | | | |
| Early Term, 6 Month Extension | XX | xx (xx.x) | xx (xx.x) |
| IV – IIIa | | xx (xx.x) | xx (xx.x) |
| IV – III vertex | | xx (xx.x) | |
| etc | | | |
| Follow-Up, 6 Month Extension | XX | xx (xx.x) | xx (xx.x) |
| IV – IIIa | | xx (xx.x) | xx (xx.x) |
| IV – III vertex | | xx (xx.x) | |
| etc | | | |

<sup>&</sup>lt;sup>a</sup> The Baseline Score → Timepoint Score combination that met the  $\ge 1$  level improvement criteria.

PROGRAMMING NOTE: Add rows for each combination that shows an improvement starting from greatest improvement and highest baseline score.

<sup>&</sup>lt;sup>b</sup> The number of patients with a non-missing score baseline and at the visit indicated. Used as denominator for percentages.

<sup>&</sup>lt;sup>c</sup> Includes early terminations or follow-ups collected during the first 26 Weeks or during the additional six months for patients opting to continue treatment in the optional six month extension. Additional rows provided to further sub-divide based on the period (1<sup>st</sup> 26 Weeks vs 6 Month Extension) and termination status (early termination vs follow-up).

Table 14.2.5
Improvement from Baseline in Sinclair Scale in Females
Safety Population

| Visit | = | Improved by $\geq 1$ Level | Improved by $\geq 2$ Levels |
|---|---|---|---|
| Shift Detail <sup>a</sup> | N <sup>b</sup> | n (%) | n (%) |
| V7 – Week 16 | XX | xx (xx.x) | xx (xx.x) |
| 4 - 3 | AA | XX (XX.X) | XX (XX.X) |
| 3 - 2 | | | ΛΛ (ΛΛ.Λ) |
| | | xx (xx.x) | |
| etc | | () | () |
| V10 – Week 26 | XX | xx (xx.x) | xx (xx.x) |
| 4 - 3 | | xx (xx.x) | xx (xx.x) |
| 3 - 2 | | xx (xx.x) | |
| etc | | | |
| V16 – Week 52 | XX | xx (xx.x) | xx (xx.x) |
| 4 - 3 | | xx (xx.x) | xx (xx.x) |
| 3 - 2 | | xx (xx.x) | , |
| etc | | () | |
| FU/Early Termination <sup>c</sup> | XX | xx (xx.x) | xx (xx.x) |
| 4 - 3 | | xx (xx.x) | xx (xx.x) |
| 3 - 2 | | xx (xx.x) | , |
| etc | | , | |
| Early Term, 1 <sup>st</sup> 26 Weeks | XX | xx (xx.x) | xx (xx.x) |
| 4 - 3 | | xx (xx.x) | xx (xx.x) |
| 3 - 2 | | xx (xx.x) | () |
| etc | | AA (AA.A) | |

 $<sup>^</sup>a$  The Baseline Score  $\to\!$  Timepoint Score combination that met the  $\geq 1$  level improvement criteria.

<sup>&</sup>lt;sup>b</sup> The number of patients with a non-missing score baseline and at the visit indicated. Used as denominator for percentages.

<sup>&</sup>lt;sup>c</sup> Includes early terminations or follow-ups collected during the first 26 Weeks or during the additional six months for patients opting to continue treatment in the optional six month extension. Additional rows provided to further sub-divide based on the period (1<sup>st</sup> 26 Weeks vs 6 Month Extension) and termination status (early termination vs follow-up).

Protocol: ATI-50002-AGA-201

Table 14.2.5
Improvement from Baseline in Sinclair Scale in Females
Safety Population

| Visit<br>Shift Detail <sup>a</sup> | $\mathbf{N^b}$ | Improved by $\geq 1$ Level n (%) | Improved by $\geq 2$ Levels n (%) |
|---|---|---|---|
| Fallan, Un 1st 26 Washer | | () | () |
| Follow-Up 1st 26 Weeks | XX | xx (xx.x) | xx (xx.x) |
| 4 - 3 | | xx (xx.x) | xx (xx.x) |
| 4 - 2 | | xx (xx.x) | |
| etc | | | |
| Early Term, 6 Month Extension | XX | xx (xx.x) | xx (xx.x) |
| 4 - 3 | | xx (xx.x) | xx (xx.x) |
| 4 - 2 | | xx (xx.x) | |
| etc | | | |
| Follow-Up, 6 Month Extension | XX | xx (xx.x) | xx (xx.x) |
| 4-3 | | xx (xx.x) | xx (xx.x) |
| 4 - 2 | | xx (xx.x) | , , |
| etc | | ` , | |

<sup>&</sup>lt;sup>a</sup> The Baseline Score → Timepoint Score combination that met the  $\ge 1$  level improvement criteria.

PROGRAMMING NOTE: Add rows for each combination that shows an improvement starting from greatest improvement and highest baseline score.

<sup>&</sup>lt;sup>b</sup> The number of patients with a non-missing score baseline and at the visit indicated. Used as denominator for percentages.

<sup>&</sup>lt;sup>c</sup> Includes early terminations or follow-ups collected during the first 26 Weeks or during the additional six months for patients opting to continue treatment in the optional six month extension. Additional rows provided to further sub-divide based on the period (1st 26 Weeks vs 6 Month Extension) and termination status (early termination vs follow-up).

Protocol: ATI-50002-AGA-201

Table 14.2.6 Correlation of Selected Effiacy Measures ITT Population

| Visit | Parameter →<br>↓ | Change in<br>Nonvellus Target<br>Area Hair Count | | Change in<br>Nonvellus Target<br>Average Area<br>Hair Width | Investigator<br>Global<br>Assessment | Subject Self<br>Assessment |
|---|---|---|---|---|---|---|
| V5 – Week 8 | Change in Nonvellus Target<br>Area Hair Count | Corr=1 | Corr=0.xx<br>P-Value=0.xxxx | Corr=0.xx<br>P-Value=0.xxxx | Corr=0.xx<br>P-Value=0.xxxx | Corr=0.xx<br>P-Value=0.xxxx |
| | Change in Nonvellus Target<br>Area Hair Width | | Corr=1 | Corr=0.xx<br>P-Value=0.xxxx | Corr=0.xx<br>P-Value=0.xxxx | Corr=0.xx<br>P-Value=0.xxxx |
| | Change in Nonvellus Target<br>Area Average Hair Width | | | Corr=1 | Corr=0.xx<br>P-Value=0.xxxx | Corr=0.xx<br>P-Value=0.xxxx |
| | Investigator Global<br>Assessment | | | | Corr=1 | Corr=0.xx<br>P-Value=0.xxxx |
| V7–Week 16<br>V10–Week 26<br>V16 – Week 52 | | | | | | |

**Note: Correlations are Pearson Correlations** 

Table 14.2.7 Correlation of Nonvellus Hair Count and Width Measures with Time Since Diagnosis of Androgenetic Alopecia ITT Population

| Visit | Parameter → ↓ | Time Since Diagnosis of Androgenetic Alopecia |
|---|---|---|
| V5 – Week 8 | Change in Nonvellus Target Area<br>Hair Count | Corr=0.xx<br>P-Value=0.xxxx |
| | Change in Nonvellus Target Area<br>Hair Width | Corr=0.xx<br>P-Value=0.xxxx |
| | Change in Nonvellus Target Area<br>Average Hair Width | Corr=0.xx<br>P-Value=0.xxxx |
| V7–Week 16<br>V10–Week 26<br>V16 – Week 52 | | |

**Note: Correlations are Pearson Correlations** 

Aclaris Therapeutics Inc.

Protocol: ATI-50002-AGA-201

23 Apr 2019 Statistical Analysis Plan

Table 14.3.1 Summary of Treatment-Emergent Adverse Events Safety Population

| | Female<br>(N=xx)<br>n (%) | Male<br>(N=xx)<br>n (%) | Total<br>(N=xx)<br>n (%) |
|---|---|---|---|
| Any Adverse Event | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Treatment-Related Adverse Event | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Serious Adverse Event | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Adverse Event Resulting in Study Discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) |

**n** = number of patients with treatment emergent adverse event(s).

NOTE: Patients with multiple occurrences of a preferred term are counted only once for that term.

Table 14.3.1.1

Treatment-Emergent Adverse Events by System Organ Class and Preferred Term Safety Population

| MedDRA SOC<br>Preferred Term | Female<br>(N=xx)<br>n (%) | Male<br>(N=xx)<br>n (%) | Total<br>(N=xx)<br>n (%) |
|---|---|---|---|
| Any Adverse Event | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AE Preferred Term 1 | xx (xx.x) | xx(xx.x) | xx (xx.x) |
| AE Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AE Preferred Term 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AE Preferred Term _ | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AE Preferred Term _ | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AE Preferred Term _ | xx (xx.x) | xx (xx.x) | xx (xx.x) |

n = number of patients with treatment emergent adverse event(s).

NOTE: Patients with multiple occurrences of a preferred term are counted only once for that term.

#### PROGRAMMING NOTE: to be carried out for:

Table 14.3.1.2 Treatment-Emergent Study Treatment-Related Adverse Events by System Organ Class and Preferred Term Safety Population

Table 14.3.1.3 Treatment-Emergent Adverse Events Resulting in Discontinuation of Study Treatment by System Organ Class and Preferred Term Safety Population

Table 14.3.1.4 Treatment-Emergent Serious Adverse Events by System Organ Class and Preferred Term Safety Population

**Table 14.3.1.5** Treatment-Emergent Adverse Events by Descending Order of Frequency for ATI-50002 **Safety Population** 

23 Apr 2019

| | Female<br>(N=xx) | Male<br>(N=xx) | Total<br>(N=xx) |
|---------------------|------------------|----------------|-----------------|
| referred Term | n (%) | n (%) | n (%) |
| AE Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AE Preferred Term 2 | xx (xx.x) | xx(xx.x) | xx (xx.x) |
| AE Preferred Term 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AE Preferred Term | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AE Preferred Term | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AE Preferred Term | xx (xx.x) | xx (xx.x) | xx (xx.x) |

n = number of patients with treatment emergent adverse event(s).

NOTE: Events presented in descending order of frequency (i.e. percentage of patients with the event) in the Total AT-50002 treatment group. Patients with multiple occurrences of a preferred term are counted only once for that term.

Protocol: ATI-50002-AGA-201

Table 14.3.1.6
Treatment-Emergent Adverse Events by Maximum Severity
Safety Population

| MedDRA SOC | | | Female, n (%) a | | |
|---|---|---|---|---|---|
| Preferred Term | Mild | Moderate | Severe | Missinga | Total |
| <b>Total Adverse Events</b> | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>&</sup>lt;sup>a</sup> Missing is referring to an event that has missing severity and no other event with severity provided for the same preferred term.

NOTE: If a patient had more than one adverse event within an SOC, the patient was counted in the category of greatest known severity.

If a patient had multiple occurrences of the same adverse event, the patient was counted in the category of greatest known severity.

Table 14.3.1.7 Treatment-Emergent Study Medication Related Adverse Events by Maximum Severity Safety Population

PROGAMMING NOTE: Separate pages for Female. Male and Total.

Protocol: ATI-50002-AGA-201

Table 14.3.1.8 Local Skin Reactions – Highest Grade Any Time Post-Baseline Safety Population

| | _ | Highest Severity, n (%) | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | • | | Fema | ale | | | Ma | ale | |
| Assessor | Sign | Mild | Moderate | Severe | Total | Mild | Moderate | Severe | Total |
| Any | Any | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Investigator | Any | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| _ | Erythema | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Scaling | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Dryness | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subject | Any | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| _ | Stinging/burning | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Itching | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>&</sup>lt;sup>a</sup> Percentages are based on the total number of patients safety population for the group.

NOTE: Patients are counted only once foreach sign at the highest severity grade.

Protocol: ATI-50002-AGA-201

**Table 14.3.1.8 Local Skin Reactions – Highest Grade Any Time Post-Baseline Safety Population** 

| _ | | | Highest | Severity, n ( | %) |
|---|---|---|---|---|---|
| | | | Tot | al | |
| Assessor | Sign | Mild | Moderate | Severe | Total |
| Any | Any | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Investigator | Any | xx(xx.x) | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| | Erythema | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Scaling | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Dryness | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subject | Any | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Stinging/burning | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Itching | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>&</sup>lt;sup>a</sup> Percentages are based on the total number of patients safety population for the group.

NOTE: Patients are counted only once foreach sign at the highest severity grade.

Table 14.3.1.9

Treatment-Emergent Adverse Events by System Organ Class and Preferred Term in Patients Who Discontinued in First 26 Weeks Safety Population

| MedDRA SOC<br>Preferred Term | Female<br>(N=xx)<br>n (%) | Male<br>(N=xx)<br>n (%) | Total<br>(N=xx)<br>n (%) |
|---|---|---|---|
| Any Adverse Event | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AE Preferred Term 1 | xx (xx.x) | xx(xx.x) | xx (xx.x) |
| AE Preferred Term 2 | xx (xx.x) | xx(xx.x) | xx (xx.x) |
| AE Preferred Term 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AE Preferred Term _ | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AE Preferred Term _ | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AE Preferred Term _ | xx (xx.x) | xx (xx.x) | xx (xx.x) |

n = number of patients with treatment emergent adverse event(s).

NOTE: Patients with multiple occurrences of a preferred term are counted only once for that term.

#### PROGRAMMING NOTE: to be carried out for:

Table 14.3.1.10 Treatment-Emergent Adverse Events by System Organ Class and Preferred Term in Patients Who Completed 26 Weeks and Did not Enter Six Month Extension Safety Population

Table 14.3.1.11 Treatment-Emergent Adverse Events by System Organ Class and Preferred Term in Patients Who Completed 26 Weeks and Entered Six Month Extension Safety Population

Table 14.3.2.1
Vital Signs: Systolic Blood Pressure (mmHg)
Safety Population

| Visit | | Fei | nale | M | ale | Total | |
|---|---|---|---|---|---|---|---|
| | Statistic | Value | Change | Value | Change | Value | Change |
| Baseline <sup>a</sup> | n | XX | | XX | | XX | |
| 2400 | Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| | Median | xxx.x | | XXX.X | | XXX.X | |
| | (Min, Max) | (xxx,xxx) | | (xxx,xxx) | | (xxx,xxx) | |
| V3 – Week 3 | n | XX | xx | XX | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| | (Min, Max) | (xxx,xxx) | (xxx, xxx) | (xxx, xxx) | (xxx,xxx) | (xxx, xxx) | (xxx, xxx) |
| V4 – Week 4 | n | xx | XX | XX | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XXX.X | xxx.x | XXX.X | xxx.x | xxx.x | xxx.x |
| | (Min, Max) | (xxx, xxx) | (xxx,xxx) | (xxx, xxx) | (xxx, xxx) | (xxx, xxx) | (xxx,xxx) |
| V5 – Week 8 | n | xx | XX | XX | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x |
| | (Min, Max) | (xxx,xxx) | (xxx,xxx) | (xxx, xxx) | (xxx,xxx) | (xxx, xxx) | (xxx, xxx) |
| V6 – Week 12 | n | XX | XX | XX | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x |
| | (Min, Max) | (xxx, xxx) | (xxx, xxx) | (xxx, xxx) | (xxx, xxx) | (xxx, xxx) | (xxx, xxx) |

<sup>&</sup>lt;sup>a</sup> Baseline is selected as the last measurement prior to the first application of study medication.

Program: XYZ.SAS

<sup>&</sup>lt;sup>b</sup> Includes early terminations or follow-ups collected during the first 26 weeks or during the additional six months for patients opting to continue treatment in the optional six month extension.

23 Apr 2019 Statistical Analysis Plan

Table 14.3.2.1
Vital Signs: Systolic Blood Pressure (mmHg)
Safety Population

| Visit | | Fe | male | M | ale | Total | |
|---|---|---|---|---|---|---|---|
| | Statistic | Value | Change | Value | Change | Value | Change |
| V7 – Week 16 | n | XX | XX | XX | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XXX.X | xxx.x | xxx.x | xxx.x | XXX.X | XXX.X |
| | (Min, Max) | (xxx,xxx) | (xxx,xxx) | (xxx, xxx) | (xxx, xxx) | (xxx, xxx) | (xxx, xxx) |
| V8 – Week 20 | n | XX | XX | XX | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x |
| | (Min, Max) | (xxx,xxx) | (xxx,xxx) | (xxx, xxx) | (xxx,xxx) | (xxx, xxx) | (xxx, xxx) |
| V9 – Week 24 | n | XX | XX | XX | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x |
| | (Min, Max) | (xxx,xxx) | (xxx,xxx) | (xxx,xxx) | (xxx,xxx) | (xxx, xxx) | (xxx, xxx) |
| V10 – Week 26 | n | XX | XX | XX | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x |
| | (Min, Max) | (xxx,xxx) | (xxx,xxx) | (xxx, xxx) | (xxx,xxx) | (xxx, xxx) | (xxx, xxx) |
| V10 – Week 26 | n | XX | XX | XX | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x |
| | (Min, Max) | (xxx,xxx) | (xxx,xxx) | (xxx,xxx) | (xxx,xxx) | (xxx, xxx) | (xxx,xxx) |

<sup>&</sup>lt;sup>a</sup> Baseline is selected as the last measurement prior to the first application of study medication.

<sup>&</sup>lt;sup>b</sup> Includes early terminations or follow-ups collected during the first 26 weeks or during the additional six months for patients opting to continue treatment in the optional six month extension.

23 Apr 2019 Statistical Analysis Plan

Table 14.3.2.1
Vital Signs: Systolic Blood Pressure (mmHg)
Safety Population

| Visit | | Fe | male | M | ale | Total | |
|---|---|---|---|---|---|---|---|
| | Statistic | Value | Change | Value | Change | Value | Change |
| V10 – Week 26 | n | XX | XX | XX | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XXX.X | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x |
| | (Min, Max) | (xxx,xxx) | (xxx,xxx) | (xxx, xxx) | (xxx, xxx) | (xxx, xxx) | (xxx, xxx) |
| V11 – Week 30 | n | XX | XX | XX | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x |
| | (Min, Max) | (xxx,xxx) | (xxx,xxx) | (xxx,xxx) | (xxx,xxx) | (xxx, xxx) | (xxx, xxx) |
| V12 – Week 35 | n | XX | XX | XX | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x |
| | (Min, Max) | (xxx,xxx) | (xxx,xxx) | (xxx, xxx) | (xxx, xxx) | (xxx, xxx) | (xxx, xxx) |
| V13 – Week 39 | n | xx | XX | XX | xx | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x |
| | (Min, Max) | (xxx,xxx) | (xxx,xxx) | (xxx,xxx) | (xxx,xxx) | (xxx, xxx) | (xxx, xxx) |
| V14 –Week 44 | n | XX | XX | XX | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x |
| | (Min, Max) | (xxx,xxx) | (xxx,xxx) | (xxx,xxx) | (xxx,xxx) | (xxx,xxx) | (xxx,xxx) |

<sup>&</sup>lt;sup>a</sup> Baseline is selected as the last measurement prior to the first application of study medication.

<sup>&</sup>lt;sup>b</sup> Includes early terminations or follow-ups collected during the first 26 weeks or during the additional six months for patients opting to continue treatment in the optional six month extension.

23 Apr 2019 Statistical Analysis Plan

Table 14.3.2.1
Vital Signs: Systolic Blood Pressure (mmHg)
Safety Population

| | | Fe | Female | | Male | | tal |
|---|---|---|---|---|---|---|---|
| Visit | Statistic | Value | Change | Value | Change | Value | Change |
| V15 – Week 48 | n | XX | XX | XX | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| | (Min, Max) | (xxx,xxx) | (xxx,xxx) | (xxx,xxx) | (xxx,xxx) | (xxx,xxx) | (xxx, xxx) |
| V16 – Week 52 | n | xx | XX | XX | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| | (Min, Max) | (xxx, xxx) | (xxx,xxx) | (xxx,xxx) | (xxx,xxx) | (xxx, xxx) | (xxx, xxx) |
| FU/Early Termination <sup>b</sup> | n | XX | XX | XX | XX | XX | XX |
| v | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x |
| | (Min, Max) | (xxx, xxx) | (xxx,xxx) | (xxx,xxx) | (xxx, xxx) | (xxx, xxx) | (xxx,xxx) |

<sup>&</sup>lt;sup>a</sup> Baseline is selected as the last measurement prior to the first application of study medication.

<sup>&</sup>lt;sup>b</sup> Includes early terminations or follow-ups collected during the first 26 weeks or during the additional six months for patients opting to continue treatment in the optional six month extension.
Aclaris Therapeutics Inc. 23 Apr 2019
Protocol: ATI-50002-AGA-201 Statistical Analysis Plan

### **PROGRAMMING NOTE:** to be repeated for the following:

| <b>Table 14.3.2.2</b> | Vital Signs | Diastolic Blood Pressure | (mmHg) Safety Population |
|---|---|---|---|
| 1 adic 14.5.4.4 | vitai bigiis. | Diastone Dioou i ressure | (miming) Saicty i opulation |

Table 14.3.2.3 Vital Signs: Heart Rate (bpm) Safety Population
Table 14.3.2.4 Vital Signs: Respiratory Rate (bpm) Safety Population
Table 14.3.2.5 Vital Signs: Temperature (Degrees C) Safety Population

23 Apr 2019 Statistical Analysis Plan

Table 14.3.3
ECG Interpretation: Shift from Baseline to Worst Assessment Post Baseline
Safety Population

| Group | Worst Post-Baseline Interpretation, n (%) | | | | |
|---|---|---|---|---|---|
| <b>Baseline Interpretation</b> | Normal | Abnormal, NCS | Abnormal, CS | Missing | Total |
| Female (Na=xx) | | | | | |
| Normal | xx(xx.x) | xx (xx.x) | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal, NCS | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal, CS | xx (xx.x) | xx (xx.x) | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Male (Na=xx) | | | | | |
| Normal | xx(xx.x) | xx (xx.x) | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal, NCS | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal, CS | xx(xx.x) | xx (xx.x) | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | xx(xx.x) | xx (xx.x) | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| Total | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total (Na=xx) | | | | | |
| Normal | xx(xx.x) | xx (xx.x) | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal, NCS | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal, CS | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>&</sup>lt;sup>a</sup> The number of all patients in the safety population for the group.

Note: The worst assessment post baseline includes any unscheduled assessment(s) as well the post-treatment assessment.

Aclaris Therapeutics Inc. 23 Apr 2019
Protocol: ATI-50002-AGA-201 Statistical Analysis Plan

PROGRAMMING NOTE: The following tables use for the format of the vital sign mean and mean change tables. Timepoints Baseline, V5 – Week 8, V7 – Week 16, V9 – Week 24, V10 – Week 26, V13 – Week 39, V14 – Week 44, V16 – Week 52, FU/Early Termination.

Table 14.3.4.1 Descriptive Statistics for Chemistry Parameters Safety Population
Table 14.3.4.2 Descriptive Statistics for Hematology Parameters Safety Population
Descriptive Statistics for Hormone Parameters Safety Population

23 Apr 2019 Statistical Analysis Plan

Table 14.3.5

Number and Percent of Patients Meeting Criteria for Hepatobiliary Laboratory Abnormalities
Safety Population

| Safety ropulation | Female | Male | Total |
|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) |
| Criteria | n (%) | n (%) | n (%) |
| >3xULN ALT or AST <sup>a</sup> | x (x.x) | x (x.x) | x (x.x) |
| >3xULN ALT | x(x.x) | x(x.x) | x(x.x) |
| >3xULN AST | x(x.x) | x(x.x) | x(x.x) |
| >5xULN ALT or AST <sup>a</sup> | x (x.x) | x (x.x) | x (x.x) |
| >5xULN ALT | x(x.x) | x(x.x) | x(x.x) |
| >5xULN AST | x(x.x) | x(x.x) | x(x.x) |
| >10xULN ALT or AST <sup>a</sup> | x (x.x) | x (x.x) | x (x.x) |
| >10xULN ALT | x(x.x) | x(x.x) | x(x.x) |
| >10xULN AST | x(x.x) | x(x.x) | x(x.x) |
| >20xULN ALT or AST <sup>a</sup> | x (x.x) | x (x.x) | x (x.x) |
| >20xULN ALT | x(x.x) | x(x.x) | x(x.x) |
| >20xULN AST | x(x.x) | x(x.x) | x(x.x) |
| Elevation of Bilirubin | | | |
| >1.5 xULN | x(x.x) | x(x.x) | x(x.x) |
| >2xULN | x(x.x) | x(x.x) | x(x.x) |
| >1.5xULN Alk Phos | x(x.x) | x(x.x) | x(x.x) |
| Elevation of AT <sup>b</sup> and Bilirubin | | | |
| >3xULN AT and >1.5xULN Bilirubin | x(x.x) | x(x.x) | x(x.x) |
| >3xULN AT and >2xULN Bilirubin | x(x.x) | x(x.x) | x(x.x) |
| >3xULN AT and >=2xULN Bilirubin and Alkaline Phosphatase <2xULN or missing | x(x.x) | x(x.x) | x(x.x) |

<sup>&</sup>lt;sup>a</sup> Patients with both ALT and AST abnormalities for the same lab draw (same date and time) are counted as one event.

PROGRAMMING NOTE: It is intentional that the last criterion has '=' added to the bilirubin threshold – to match exactly FDA Guidance doc

<sup>&</sup>lt;sup>b</sup> AT = aminotransferase. Either AST or ALT (or both) elevated.

23 Apr 2019 Statistical Analysis Plan

Table 14.3.6 Number and Percent of Patients Meeting Laboratory Criteria for Potential Renal Impairment Safety Population

| Criteria | Female (N=xx) n (%) | Male<br>(N=xx)<br>n (%) | Total<br>(N=xx)<br>n (%) |
|---|---|---|---|
| Change from Baseline ≥ 0.5 mg/dL | x (x.x) | x (x.x) | x (x.x) |
| >1.5xULN Creatinine | x(x.x) | x(x.x) | x(x.x) |
| EITHER Change from Baseline >=0.5 mg/dL or >1.5xULN Creatinine | x(x.x) | x(x.x) | x(x.x) |
| BOTH Change from Baseline >= 0.5 mg/dL and >1.5xULN Creatinine | x(x.x) | x(x.x) | x(x.x) |

Figure 14.1
Association of Selected Efficacy Measures with Fit Linear Regression Line
ITT Population: Visit = V5 Week 8



#### Reperat for:

| Figure 14.2 | Association of Selected Efficacy Measures with Fit Linear Regression Line, ITT Population: Visit=V7 Week 16 |
|---|---|
| Figure 14.3 | Association of Selected Efficacy Measures with Fit Linear Regression Line, ITT Population: Visit=V10 Week 26 |
| Figure 14.4 | Association of Selected Efficacy Measures with Fit Linear Regression Line, ITT Population: Visit=V16 Week 52 |

For the following plot change in averge hair wdth (vertical) vs Investigaor Global Assessment [4 figures – All timepoints on page]. Indicate timepoint at top of each of the visits. Separate color for males and females and linear regression line as per figure 14.1.Add Foonote: Note Lines represent fit linear regression line.

Figure 14.5 Association of Change in Nonvellus Target Area Average Hair Width with Investigator Global Assessment, ITT Population

For the following plot change in averge hair wdth (vertical) vs Subject Self Assessment [4 figures – All timepoints on page] Indicate timepoint at top of each of the visits. Separate color for males and females and linear regression line as per figure 14.1.Add Foonote: Note Lines represent fit linear regression line.

Figure 14.6 Association of Change in Nonvellus Target Area Average Hair Width with Subject Self Assessment, ITT Population

For the following plot change nonvellus target area hair count (vertical), change nonvellus target area hair width (vertical) and change nonvellus target area average hair width (vertical), vs time since diagnosis of androgenetic alopecia [4 figures on page – all timepoints on page] Indicate timepoint at top of each of the visits. Separate color for males and females and linear regression line as per figure 14.1.Add Foonote: Note Lines represent fit linear regression line.

| Figure 14.7 | Association of Change in Nonvellus Target Area Hair Count with Time Since Diagnosis of Androgenetic Alopecia, ITT Population |
|---|---|
| Figure 14.8 | Association of Change in Nonvellus Target Area Hair Width with Time Since Diagnosis of Androgenetic Alopecia, ITT Population |
| Figure 14.9 | Association of Change in Nonvellus Target AreaAverage Hair Width with Time Since Diagnosis of Androgenetic Alopecia, ITT |
| Population | |

23 Apr 2019 Statistical Analysis Plan

Protocol: ATI-50002-AGA-201

# Appendix 16.2.1.1 Disposition

### Group: Female, Male

| <u>Patient</u> | Date of<br>Last<br>Application <sup>a</sup> | Date of DC/<br>Completion | Days from Last<br>Application <sup>b</sup> | | Reason DC from Study | Period of Study<br>Discontinuation/<br>Completion |
|---|---|---|---|---|---|---|
| xx-xxx | mmdddyy | mmdddyy | XX | xx | Adverse Event/SAE: list AE, link by AE number Protocol Violation Lost to Follow-Up Withdrew Consent Pregnancy Other: specify Completed | First 26 Weeks<br>6 Month Extension |

<sup>&</sup>lt;sup>a</sup> Date of last dose of application of study medication.

**NOTE: DC=Discontinued.** 

b DC date/Completion Date- date last application +1.

<sup>&</sup>lt;sup>c</sup> DC date/ Completion Date – date of first application of study medication +1.

23 Apr 2019 Statistical Analysis Plan

Protocol: ATI-50002-AGA-201

# Appendix 16.2.1.2 Demographics

| Patient | Age <sup>a</sup><br>(Years) | Gender | Race | Ethnicity | Fitzpatrick<br>Skin Type | Height <sup>b</sup><br>(inches) | Weight <sup>l</sup><br>(lbs) |
|---|---|---|---|---|---|---|---|
| xx-xxx | XX | Male<br>Female | Caucasian/White Black Asian/Oriental American Indian or Alaska Native Native Hawaiian or Pacific Islander Other - specify | Hispanic/Latino<br>Not Hispanic/Latino<br>Not Willing to Provide | 1,2,3,4,5,6 | xx.x | xxx<br>xxx.x |

<sup>&</sup>lt;sup>a</sup> At Date of signed informed consent.

<sup>&</sup>lt;sup>b</sup> FromV-2 Day 1 vitals page.

23 Apr 2019 Statistical Analysis Plan Protocol: ATI-50002-AGA-201

#### **Appendix 16.2.1.3** History of Androgenetic Alopecia: Diagnosis and Prior Treatment and Therapies

Group: Female, Male

| Patient | Onset Date of Diagnosis | Years Since<br>Diagnosis <sup>a</sup> | Prior Treatment/<br>Therapy Type | Treatment or Therapy<br>Coded/Verbatim | Start Date/<br>Stop Date | Start Day <sup>b</sup> / Stop Day <sup>b</sup> |
|---|---|---|---|---|---|---|
| xx-xxx | ddmmmyyyy | XX.X | Pharmaceutical | Minoxidil/ | 01Jan2018 | 55 |
| | | | | Rogaine/ | 03Jan2018 | 57 |
| | | | Pharmaceutical | Finasteride/ | 01Jan2018 | 55 |
| | | | | Propecia | 03Jan2018 | 57 |
| | | | Device | Coded term/<br>verbatim | | |
| | | | Other | Coded term/<br>verbatim | | |

NOTE: Date of Diagnosis from medical history page of CRF

PROGRAMMING NOTE: Will need to review prior treatment and therapies to assign "Type" i.e. "Pharmaceutical", "Device" and "other"

<sup>&</sup>lt;sup>a</sup> (Date of Diagnosis - Date of first application of study medication) / 365.

<sup>&</sup>lt;sup>b</sup> Start date – date of first application of study medication

23 Apr 2019 Statistical Analysis Plan

Protocol: ATI-50002-AGA-201

#### Appendix 16.2.1.4 Medical History

Group: Female, Male

| Patient | Body System | Diagnosis | Onset<br>Date (Study Day <sup>a</sup> ) | Resolution Date (Study Day <sup>a</sup> ) | Ongoing at Time of Randomization? |
|---|---|---|---|---|---|
| xx-xxx | Skin | Free Text | ddmmmyyyy (xx) | ddmmmyyyy (xx) | Yes |
| | Central nervous system | | , | | |
| | Ophthalmologic | | | | |
| | Ear, nose, throat | | | | |
| | Respiratory | | | | |
| | Gastrointestinal | | | | |
| | Hepatic | | | | |
| | Renal | | | | |
| | Cardiovascular | | | | |
| | Hematologic | | | | |
| | Genitourinary | | | | |
| | Endocrine/Lymphatic<br>Musculoskeletal | | | | |
| | Systemic Infection | | | | |
| | Drug Allergy | | | | |
| | Substance Abuse | | | | |
| | Psychiatric Psychiatric | | | | |
| | Other | | | | |

<sup>&</sup>lt;sup>a</sup> Study Day = Start/stop date - date of first application of study medication.

PROGRAMMING NOTE: List dates as entered - i.e., display partial dates. Imputed dates in database are used to calculate study day. If patient has no entries, put "None" under Body System.

23 Apr 2019 Statistical Analysis Plan

Protocol: ATI-50002-AGA-201

## Appendix 16.2.1.5 Prior and Concomitant Therapies

Group: Female, Male

| Patient | WHO ATC Level III/<br>WHO Preferred Term/<br>Verbatim Term | Dose (unit)<br>[Route] Frequency | Study Period(s)<br>in Which<br>Received <sup>a</sup> | | Start Day <sup>b</sup> / Stop Day <sup>b</sup> | Indication | Associated<br>with AE<br>(AE#) |
|---|---|---|---|---|---|---|---|
| | | xx (mg) [oral] QD | P<br>O<br>F<br>P,O<br>O,F<br>P,O,F | 01Jan2018<br>03Jan2018 | | Free Text | No<br>Yes (xx) |
| | | | 1,0,1 | Note: if "ongoing", put "ongoing" under Stop Date | | | |

**NOTE:** -= data not available

<sup>&</sup>lt;sup>a</sup> P = Prior medication; O = Treatment Period; F=Post-Therapy

b Start date – date of first application of study medication (+1 if ≥ first application of study medication).

23 Apr 2019 Statistical Analysis Plan

Protocol: ATI-50002-AGA-201

#### Appendix 16.2.1.6 ATI-50002 Accountability

| | | | Dispensed | | | | | V | olume |
|---|---|---|---|---|---|---|---|---|---|
| Patient | Date<br>Dispensed | Study<br>Day <sup>a</sup><br>Dispensed | Bottle Weight Date (gm) Collected | | Study Day <sup>a</sup><br>Collected | Collected<br>Bottle Weight<br>(gm) | Amount -<br>Used <sup>b</sup><br>(gm) | (mL) <sup>c</sup> | Volume (mL) Per<br>Application <sup>c</sup> |
| xx-xxx | ddmmmyyyy | XX | XX | ddmmmyyyy | XX | XX | XX | XX | |
| | ddmmmyyyy | | XX | ddmmmyyyy | XX | XX | XX | XX | |
| | ddmmmyyyy | XX | XX | ddmmmyyyy | XX | XX | XX | XX | |
| | | | | | | TOTAL: | XX | XXX | XX.X |

<sup>&</sup>lt;sup>a</sup> Dispensed Date (or Collection Date) – Date first Application +1.

<sup>&</sup>lt;sup>b</sup> Weight dispensed – Weight collected (returned).

<sup>&</sup>lt;sup>c</sup> The density of study agent is 1 g/mL which is used to convert differences in bottle weights between dispensed and returned (ie weight of study agent used) to mLs.

23 Apr 2019 Statistical Analysis Plan

Protocol: ATI-50002-AGA-201

# Appendix 16.2.1.7 ATI-50002 Accountability Comments

| | Date | Study Day <sup>a</sup><br>Dispensed | Date | Study<br>Day <sup>a</sup> | |
|---|---|---|---|---|---|
| Patient | Dispensed | | Collected | Collected | Comment |
| xx-xxx | ddmmmyyyy | XX | ddmmmyyyy | XX | Free Text |
| | ddmmmyyyy | XX | ddmmmyyyy | XX | |
| | ddmmmyyyy | XX | ddmmmyyyy | XX | |

<sup>&</sup>lt;sup>a</sup> Dispensed Date (or Collection Date) – Date first Application +1.

23 Apr 2019 Statistical Analysis Plan

Protocol: ATI-50002-AGA-201

# Appendix 16.2.1.8 ATI-50002 Application Changes and Missed Doses

| Patient | Application Frequency<br>Started | Study Day <sup>a</sup><br>Dispensed | Application Frequency<br>Ended | Study Day <sup>a</sup><br>Collected | Applications/Day |
|---|---|---|---|---|---|
| XX-XXX | ddmmmyyyy | XX | ddmmmyyyy | XX | XX |
| | ddmmmyyyy | XX | ddmmmyyyy | XX | XX |
| | ddmmmyyyy | XX | ddmmmyyyy | XX | XX |

<sup>&</sup>lt;sup>a</sup> Dispensed Date (or Collection Date) – Date first Application +1.

23 Apr 2019 Statistical Analysis Plan

Protocol: ATI-50002-AGA-201

# Appendix 16.2.1.9

### Group: Female, Male

| Patient | Inclusion Criteria Not Met | Exclusion Criteria Not Met |
|---------|----------------------------|----------------------------|
| | 1,213 | None |
| | None | 1,216 |

**Eligibility Criteria** 

| Aclaris Therapeutics Inc. | 23 Apr 2019 |
|-----------------------------|---------------------------|
| Protocol: ATI-50002-AGA-201 | Statistical Analysis Plan |

### Appendix 16.2.1.10 Protocol Violations

| Group: Fe | male, Male |
|-----------|------------|
| Patient | Violation |

23 Apr 2019 Statistical Analysis Plan

Appendix 16.2.2.1
Target Area Hair Count and Width

| Group: Fem | Group: Female, Male | | | | |
|---|---|---|---|---|---|
| Patient | Visit | Assessment Date | Study Day <sup>a</sup> | TAHC<br>(hairs/cm²) | TAHW<br>(cm) |
| xx-xxx | V2 – Day 1 | ddmmmyyyy | XX | xxx | xxx |
| | V5 – Week 8 | ddmmmyyyy | XX | XXX | XXX |
| | V7 – Week 16 | ddmmmyyyy | XX | XXX | XXX |
| | V10 – Week 26 | ddmmmyyyy | XX | XXX | XXX |
| | V16 – Week 52 | ddmmmyyyy | XX | XXX | XXX |

<sup>&</sup>lt;sup>a</sup> Assessment date – date of first application of study medication (+1 if ≥ first application of study medication).

23 Apr 2019 Statistical Analysis Plan

Protocol: ATI-50002-AGA-201

#### Appendix 16.2.2.2 Investigator and Subject Global Assessments

| Patient | Visit | Assessment<br>Date | Study<br>Day <sup>a</sup> | Investigator<br>Global<br>Assessment <sup>b</sup> | Subject<br>Global<br>Assessment <sup>t</sup> |
|---|---|---|---|---|---|
| xx-xxx | V5 – Week 8 | ddmmmyyyy | XX | -3 | -3 |
| AA AAA | V7 – Week 16 | ddmmmyyyy | XX | -2 | -2 |
| | V10 – Week 26 | ddmmmyyyy | XX | -1 | -1 |
| | V13 – Week 39 | ddmmmyyyy | XX | 0 | 0 |
| | V16 – Week 52 | ddmmmyyyy | XX | 1 | 1 |
| | Early Term 1st 26 Weeks | ddmmmyyyy | XX | 2 | 2 |
| | Follow-Up 1st 26 Weeks | 3333 | | 3 | 3 |
| | Early Term 6 Month Extension | | | | |
| | Follow-Up 6 Month Extension | | | | |

Programming note: Differentiation between Early term and Follow-up is based on the availability of V10 (1st 26 Weeks) or V16 (patients entering extension) data for ANY data (not just global assessments). If a patient does not enter the extension and had no data collected for V10 and had discontinued the trial the follow-up is considered "Early Term 1st 26 Weeks". If they had V10 and did not enter the extension then it's "Follow-Up 6 Month Extension". Similarly for those entering extension, those without a V16 who discontinued the study are assigned "Early Term 6 Month Extension" and those with V16 are assigned to "Follow-Up 6 Month Extension".

<sup>&</sup>lt;sup>a</sup> Assessment date – date of first application of study medication (+1 if ≥ first application of study medication).

b -3: Greatly decreased hair growth; -2: Moderately decreased hair growth; -1: Slightly decreased hair growth; 0: No Change; +1: Slightly increased hair growth; +2: Moderately increased hair growth; +3: Greatly increased hair growth.

#### Appendix 16.2.2.3 Norwood-Hamilton Scale in Males

| Patient | Visit | Assessment<br>Date | Study<br>Day <sup>a</sup> | N-H Score | Improvement<br>from Baseline<br>(Yes/No) <sup>c</sup> |
|---|---|---|---|---|---|
| VV VVV | V1 Caraanina | ddmmmraaa | WW | I | Yes/No |
| XX-XXX | V1 - Screening<br>V2 – Day 1 | ddmmmyyyy | XX<br>XX | $\Pi_{\mathrm{p}}$ | I ES/INO |
| | V2 – Day 1<br>V7 – Week 16 | ddmmmyyyy<br>ddmmmyyyy | XX | II<br>IIa | |
| | V10 – Week 16<br>V10 – Week 26 | ddmmmyyyy | | IIa<br>III | |
| | V16 – Week 20<br>V16 – Week 52 | | XX | IIIa | |
| | | ddmmmyyyy | XX | | |
| | Early Term 1 <sup>st</sup> 26 Weeks<br>Follow-Up 1 <sup>st</sup> 26 Weeks | ddmmmyyyy | XX | III Vertex<br>IV | |
| | * | | | IV<br>IVa | |
| | Early Term 6 Month Extension | | | Iva<br>V | |
| | Follow-Up 6 Month Extension | | | · | |
| | | | | Va<br>VI | |
| | | | | VI<br>VII | |

<sup>&</sup>lt;sup>a</sup> Assessment date – date of first application of study medication (+1 if ≥ first application of study medication).

Programming note: Differentiation between Early term and Follow-up is based on the availability of V10 (1st 26 Weeks) or V16 (patients entering extension) data for ANY data (not just Norwood-Hamilton). If a patient does not enter the extension and had no data collected for V10 and had discontinued the trial the follow-up is considered "Early Term 1st 26 Weeks". If they had V10 and did not enter the extension then it's "Follow-Up 1st 26 Weeks". Similarly for those entering extension, those without a V16 who discontinued the study are assigned "Early Term 6 Month Extension" and those with V16 are assigned to "Follow-Up 6 Month Extension".

<sup>&</sup>lt;sup>b</sup> Used as baseline for analysis.

<sup>&</sup>lt;sup>c</sup> Yes – score improved by ≥1 level including shifts in "sub-level" (e.g. IIIa to III is considered a 1 level improvement).

Appendix 16.2.2.4 Sinclair Scale in Females

| Patient | Visit | Assessment<br>Date | Study<br>Day <sup>a</sup> | Sinclair Score | Improvement<br>from Baseline<br>(Yes/No) |
|---|---|---|---|---|---|
| xx-xxx | V1 - Screening | ddmmmyyyy | XX | 1 | Yes/No |
| | V2 – Day 1 | ddmmmyyyy | XX | 2 <sup>b</sup> | |
| | V7 – Week 16 | ddmmmyyyy | XX | 3 | |
| | V10 – Week 26 | ddmmmyyyy | XX | 4 | |
| | V16 – Week 52 | ddmmmyyyy | XX | 5 | |
| | Early Term 1 <sup>st</sup> 26 Weeks<br>Follow-Up 1 <sup>st</sup> 26 Weeks<br>Early Term 6 Month Extension<br>Follow-Up 6 Month Extension | ddmmmyyyy | XX | | |

Programming note: Differentiation between Early term and Follow-up is based on the availability of V10 (1st 26 Weeks) or V16 (patients entering extension) data for ANY data (not just Sinclair score). If a patient does not enter the extension and had no data collected for V10 and had discontinued the trial the follow-up is considered "Early Term 1st 26 Weeks". If they had V10 and did not enter the extension then it's "Follow-Up 1st 26 Weeks". Similarly for those entering extension, those without a V16 who discontinued the study are assigned "Early Term 6 Month Extension" and those with V16 are assigned to "Follow-Up 6 Month Extension".

<sup>&</sup>lt;sup>a</sup> Assessment date – date of first application of study medication (+1 if ≥ first application of study medication).

<sup>&</sup>lt;sup>b</sup> Used as baseline for analysis.

23 Apr 2019 Statistical Analysis Plan Protocol: ATI-50002-AGA-201

#### **Appendix 16.2.3.1** All Adverse Events

**Group: Female, Male** 

| Patient | MedDRA SOC/<br>MedDRA Preferred Term/<br>CRF Verbatim Term (AE No.) | Onset Study Day <sup>a</sup><br>Resolution Study Day <sup>b</sup><br>Duration (Days) <sup>c</sup> | Onset Date/<br>Stop Date<br>Cutaneous AE? | Relationship/<br>Action Taken/<br>Therapy Required | Serious/<br>Severity/<br>Outcome |
|---|---|---|---|---|---|
| 501-01 | Cardiovascular System / | 62 | 01Sep12 | Related | Yes/No |
| | Bradycardia / | 64 | | Not Related | |
| | Slow Heart Rate (xx) <sup>d</sup> | 3 | 03Sep12 | | Mild/Moderate/Severe |
| | | | Ongoing | Dose not changed | |
| | | | 0 0 | Dose Reduced | Recoverd/Resolved |
| | | | Yes (Scalp), | Dose Interrupted | Not Recovered/Resolved |
| | | | Yes (not Scalp), | Drug Withdrawn | Recovered/Resolved w/ Seq. |
| | | | No | Unknown | Fatal<br>Unknown |
| | | | | Yes/No | |

<sup>&</sup>lt;sup>a</sup> AE onset date – date of first application of study medication (+1 if ≥ first application).

### PROGRAMMING NOTES: Sort by group, patient, onset date, SOC and PREF term. Display partial dates as entered in raw data. Use derived dates for study day and duration

**Appendix 16.2.3.2 Serious Adverse Events** 

**Adverse Events Resulting in Discontinuation of Study Treatment Appendix 16.2.3.3** 

**Appendix 16.2.3.4 Adverse Events Resulting in Outcome of Death** 

<sup>&</sup>lt;sup>b</sup> AE resolution date – date of first application of study medication (+1 if ≥ first application).

<sup>&</sup>lt;sup>c</sup> Resolution Date – Onset Date +1

<sup>&</sup>lt;sup>d</sup> Not treatment emergent = Onset either prior to the first application or > 30 days after the last application of study medication.

23 Apr 2019 Statistical Analysis Plan

Protocol: ATI-50002-AGA-201

#### Appendix 16.2.3.5 Local Skin Reactions

| Patient | Visit | Assessment<br>Date | Study<br>Day <sup>a</sup> | Assessor | Sign <sup>b</sup> | Grade |
|---|---|---|---|---|---|---|
| | V2 – Day 1 | ddmmmyyyy | 1 | Investigator | Erythema | 1 |
| | • | | | - | Scaling | 2 |
| | | | | | Dryness | 3 |
| | | | | Subject | Stinging/burning | |
| | | | | • | Itching | |
| | | | | Investigator | NO SIGN GRADED >0 | |
| | | | | Subject/Legal Guardian | NO SIGN GRADED >0 | |
| | V3 – Week 3 | ddmmmyyyy | 21 | | | |

<sup>&</sup>lt;sup>a</sup> Assessment Date – Date first Application +1.

<sup>&</sup>lt;sup>b</sup> Only signs with grade > 0 are displayed. Within assessor, if all signs were grade 0 (or not done) appear as "NO SIGN GRADED > 0".

23 Apr 2019 Statistical Analysis Plan

Protocol: ATI-50002-AGA-201

#### Appendix 16.2.3.6 Physical Exam

Group: Female, Male

| Patient | Assessment<br>Date | Visit | Study<br>Day <sup>a</sup> | Body<br>System | Finding <sup>b</sup> | Description of Finding |
|---|---|---|---|---|---|---|
| xx-xxx | ddmmmyyyy | V1 – Screening<br>ET/Follow-Up | XX | | Normal, no findings | |
| | | 1 | | Body System a<br>Body System b | Abnormal, CS<br>Abnormal, NCS | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

NOTE: Listing includes only lists body systems that were assessed with Abnormalities. Patients with only "normal" findings are listed as "Normal, no findings" (can have some body systems "not done" so long as those that were assessed are all "normal". Not done are not listed.)

<sup>&</sup>lt;sup>a</sup> Assessment Date – Date of First Application (+1 if ≥ first application of study medication).

<sup>&</sup>lt;sup>b</sup> CS = Clinically Significant; NCS = Not Clinically Significant

23 Apr 2019 Statistical Analysis Plan

Protocol: ATI-50002-AGA-201

#### Appendix 16.2.3.7 Vital Signs

| | | | | | _ | Blood Pressure |
|---|---|---|---|---|---|---|
| D-4'4 | ¥7°*4 | C4 J D3 | Heart Rate | Respiratory Rate | Temperature | Systolic / Diastolic |
| <b>Patient</b> | Visit | Study Day <sup>a</sup> | (bpm) | (bpm) | (Degrees C) | (mmHg) |
| xx-xxx | V1 – Screening | XX | XXX | XX | XX | xxx / xxx |
| | V2 – Day 1 | | | | | |
| | V3 – Week 3 | | | | | |
| | V4 – Week 4 | | | | | |
| | V5 – Week 8 | | | | | |
| | V6 – Week 12 | | | | | |
| | V7 – Week 16 | | | | | |
| | V8 – Week 20 | | | | | |
| | V9 – Week 24 | | | | | |
| | V10 – Week 26 | | | | | |
| | ET/Follow-Up | | | | | |
| | V11 – Week 30 | | | | | |
| | V12 – Week 35 | | | | | |
| | V13 – Week 39 | | | | | |
| | V14 – Week 44 | | | | | |
| | V15 – Week 48 | | | | | |
| | V15 – Week 52 | | | | | |
| | Follow-Up/ Early Termination <sup>b</sup> | | | | | |

<sup>&</sup>lt;sup>a</sup> Assessment Date – Date of First Application (+1 if ≥ first application of study medication).

<sup>&</sup>lt;sup>b</sup> Includes early terminations or follow-ups collected during the first 26 Weeks or during the additional six months for patients opting to continue treatment in the optional six month extension.

23 Apr 2019 Statistical Analysis Plan

Protocol: ATI-50002-AGA-201

#### Appendix 16.2.3.8 Electrocardiogram – Evaluator Interpretation

Group: Female, Male

| Patient | Visit | Study Day <sup>a</sup> | Interpretation <sup>b</sup> | Specify – if abnormal |
|---|---|---|---|---|
| XX-XXX | | XX | Normal | |
| | | XX | Abnormal, CS | Sinus Bradycardia |
| | | XX | Abnormal, NCS | Inverted T Waves; T Wave Abnormality: Biphasic T Waves |
| | | XX | Abnormal, NCS | • • |

Programming Note: Suggestion is to list all abnormalities at a given collection be listed according to "interpretation" (ie CS and/or NCS). So if there are multiple reasons, as in the hypothetical example above for NCS, separate them by semi-colons.

<sup>&</sup>lt;sup>a</sup> Assessment Date – Date of First Application (+1 if ≥ first application of study medication).

<sup>&</sup>lt;sup>b</sup> CS = Clinically Significant; NCS = Not Clinically Significant

23 Apr 2019 Statistical Analysis Plan

Protocol: ATI-50002-AGA-201

### Appendix 16.2.3.9 Clinical Laboratory Assessments: Hematology

Group: Female, Male

| Patient | Age<br>(years) | Gender | Parameter (unit) | Visit | Study<br>Day <sup>a</sup> | Value | Normal<br>Range | | List Criteria Met, if applicable, for Hold of Study Medication |
|---|---|---|---|---|---|---|---|---|---|
| xx-xxx | 60 | Female | Hemoglobin (g/dL) | | -10<br>-1 <sup>b</sup><br>28<br>38 | XXX<br>XXX<br>XXX<br>XXX | XX.X-XX.X | L<br>H | < 8 g/dL or decrease > 2 g/dL |
| | | | Hematocrit (%) | | | | | | |

<sup>&</sup>lt;sup>a</sup> Assessment Date – Date of First Application (+1 if ≥ first application of study medication).

PROGRAMMING NOTE: Sort by group, patient, parameter, and study day. For criteria for holding study medication see protocol – Section 10.2.4.1

| | Repeat format for: |
|--------------------|--------------------------------------------------|
| Appendix 16.2.3.10 | Clinical Laboratory Assessments: Biochemistry |
| Appendix 16.2.3.11 | <b>Clinical Laboratory Assessments: Hormones</b> |

<sup>&</sup>lt;sup>b</sup> Value used for baseline.

23 Apr 2019 Statistical Analysis Plan

Protocol: ATI-50002-AGA-201

Appendix 16.2.3.12

Group: Female, Male

| Patient | Age<br>(years) | Gender | Parameter | Visit | Study<br>Day <sup>a</sup> | Value |
|---|---|---|---|---|---|---|
| | 60 | Female | Glucose | | -10<br>-1 <sup>b</sup> | Positive<br>Negative<br>Trace |
| | | | Protein<br>RBC<br>WBC<br>Urobilinogen | | XX | |

**Clinical Laboratory Assessments: Urinalysis** 

PROGRAMMING NOTES: Display parameters in alphabetical order.
Sort by group, patient, parameter, and study day.

<sup>&</sup>lt;sup>a</sup> Assessment Date – Date of First Application (+1 if ≥ first application of study medication).

<sup>&</sup>lt;sup>b</sup> Value used for baseline.

23 Apr 2019 Statistical Analysis Plan

Protocol: ATI-50002-AGA-201

## Appendix A MedDRA System Organ Class/Preferred Term and CRF Verbatim Terms

**MedDRA System Organ Class** 

**MedDRA Preferred Term** 

**CRF Verbatim Term** 

NOTE: Events coded using MedDRA Version 21.1